CLINICAL TRIAL: NCT02753127
Title: A Phase 3 Study of BBI-608 in Combination With 5-Fluorouracil, Leucovorin, Irinotecan (FOLFIRI) in Adult Patients With Previously Treated Metastatic Colorectal Cancer (CRC).
Brief Title: A Study of Napabucasin (BBI-608) in Combination With FOLFIRI in Adult Patients With Previously Treated Metastatic Colorectal Cancer
Acronym: CanStem303C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CanStem303C; BB608-303CRC (Other: Sumitomo Dainippon Pharma Oncology, Inc.); 2016-001627-31 (EudraCT Number)
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Results first posted 2022-04-26 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Neoplasms; Colonic Diseases; Digestive System Diseases; Digestive System Neoplasms; Gastrointestinal Diseases; Gastrointestinal Neoplasms; Intestinal Diseases; Intestinal Neoplasms; Neoplasms; Neoplasms by Histologic Type; Neoplasms by Site; Neoplasms, Glandular and Epithelial; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Diseases; Digestive System Diseases; Digestive System Neoplasms; Gastrointestinal Diseases; Gastrointestinal Neoplasms; Intestinal Diseases; Intestinal Neoplasms; Neoplasms; Neoplasms by Histologic Type; Neoplasms by Site; Neoplasms, Glandular and Epithelial; Rectal Diseases | interventions — napabucasin; Fluorouracil; Leucovorin; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Napabucasin plus FOLFIRI (Experimental): Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will start at least 2 hours following the first daily dose of napabucasin and will be administered every 2 weeks. Irinotecan/leucovorin infusion will follow bevacizumab infusion in selected patients to receive standard dose of bevacizumab (5 mg/kg). Irinotecan 180 mg/m^2 together with leucovorin 400 mg/m^2 will be administered intravenously, over approximately 90 minutes and 2 hours, respectively, starting on Day 1 of Cycle 1, following bevacizumab infusion or at least 2 hours following the first daily dose of napabucasin if bevacizumab is not administered. 5-FU 400 mg/m^2 bolus will be administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m^2/day (total 2400 mg/m^2) continuous infusion. This regimen will be repeated on Day 1 of every 14 day cycle.
  Interventions: Drug: Napabucasin; Drug: Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Bevacizumab
- FOLFIRI (Active Comparator): Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will be administered every 2 weeks. Irinotecan/leucovorin infusion will follow bevacizumab infusion in selected patients to receive standard dose of bevacizumab (5 mg/kg). Irinotecan 180 mg/m^2 together with leucovorin 400 mg/m^2 will be administered intravenously, over approximately 90 minutes and 2 hours, respectively, starting on Day 1 of Cycle 1, following bevacizumab infusion. 5-FU 400 mg/m^2 bolus will be administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m^2/day (total 2400 mg/m^2) continuous infusion. This regimen will be repeated on Day 1 of every 14 day cycle.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Irinotecan; Drug: Bevacizumab

INTERVENTIONS:
Drug: Napabucasin — Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 12 hours (480 mg total daily dose).
  Other Names: BBI-608; BBI608; BB608
  Arms: Napabucasin plus FOLFIRI
Drug: Fluorouracil
  Other Names: 5-FU; Carac; Efudex; Fluoroplex; Adrucil
Drug: Leucovorin
  Other Names: Folinic Acid
Drug: Irinotecan
  Other Names: Camptosar
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
This is an international multi-center, prospective, open-label, randomized, adaptive design phase 3 trial of the cancer stem cell pathway inhibitor napabucasin plus standard bi-weekly FOLFIRI versus standard bi-weekly FOLFIRI in patients with previously treated metastatic colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed consent for trial participation must be obtained from the patient appropriately in accordance with applicable ICH guidelines and local and regulatory requirements prior to the performance of any study specific procedure.
2. Must have histologically confirmed advanced CRC that is metastatic.
3. Must have failed treatment with one regimen containing a fluoropyrimidine, oxaliplatin with or without bevacizumab for metastatic disease. All patients must have received a minimum of 6 weeks of the first-line regimen that included bevacizumab (if applicable), oxaliplatin and a fluoropyrimidine in the same cycle. Treatment failure is defined as radiologic progression during or < 6 months after the last dose of first-line therapy.
4. FOLFIRI therapy is appropriate for the patient and is recommended by the Investigator.
5. Imaging investigations including CT/MRI of chest/abdomen/pelvis or other scans as necessary to document all sites of disease performed within 21 days prior to randomization. Patients with either measurable disease or non-measurable evaluable disease are eligible.
6. Must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Must be ≥ 18 years of age.
8. For male or female patient of child bearing potential: Must agree to use contraception or take measures to avoid pregnancy during the study and for 180 days for female and male patients, of the final FOLFIRI dose. Patients who receive single agent napabucasin without FOLFIRI must agree to use contraception or take measures to avoid pregnancy during the study and for 30 days for female patients and 90 days for male patients, of the final napabucasin dose.
9. Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test within 5 days prior to randomization. The minimum sensitivity of the pregnancy test must be 25 IU/L or equivalent units of HCG.
10. Must have alanine transaminase (ALT) ≤ 3 × institutional upper limit of normal (ULN) [≤ 5 × ULN in presence of liver metastases] within 14 days prior to randomization.
11. Must have hemoglobin (Hgb) ≥ 9.0 g/dL within 14 days prior to randomization. Must not have required transfusion of red blood cells within 1 week of baseline Hgb assessment.
12. Must have total bilirubin ≤ 1.5 × institutional ULN [≤ 2.0 x ULN in presence of liver metastases] within 14 days prior to randomization.
13. Must have creatinine ≤ 1.5 × institutional ULN or Creatinine Clearance > 50 ml/min (as calculated by the Cockcroft-Gault equation (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) within 14 days prior to randomization.
14. Must have absolute neutrophil count ≥ 1.5 x 10^9/L within 14 days prior to randomization.
15. Must have platelet count ≥ 100 x 10^9/L within 14 days prior to randomization. Must not have required transfusion of platelets within 1 week of baseline platelet assessment.
16. Patient must have adequate nutritional status with Body Mass Index (BMI) > 18 kg/m^2 and body weight of > 40 kg with serum albumin > 3 g/dL.
17. Other baseline laboratory evaluations, listed in Section 6.0, must be done within 14 days prior to randomization.
18. Patient must consent to provision of, and Investigator(s) must confirm access to and agree to submit a representative formalin fixed paraffin block of tumor tissue in order that the specific biomarker assays may be conducted. Submission of the tissue is to occur prior to randomization, unless approved by the Sponsor. Where local center regulations prohibit submission of blocks of tumor tissue, two 2 mm cores of tumor from the block and 10-30 unstained slides of whole sections of representative tumor tissue are preferred. Where two 2 mm cores of tumor from the block are unavailable, 10-30 unstained slides of whole sections of representative tumor tissue alone are acceptable. Where no previously resected or biopsied tumor tissue exists or is available, on the approval of the Sponsor/designated CRO, the patient may still be considered eligible for the study.
19. Patient must consent to provision of a sample of blood in order that the specific correlative marker assays may be conducted.
20. Patients must be accessible for treatment and follow-up. Patients registered on this trial must receive protocol treatment and be followed at the participating center. This implies there must be reasonable geographical limits placed on patients being considered for this trial. Investigators must ensure that the patients randomized on this trial will be available for complete documentation of the treatment, response assessment, adverse events, and follow-up.
21. Protocol treatment is to begin within 2 calendar days of patient randomization.
22. The patient is not receiving therapy in a concurrent clinical study and the patient agrees not to participate in other interventional clinical studies during their participation in this trial while on study treatment. Patients participating in surveys or observational studies are eligible to participate in this study.

Exclusion Criteria:

1. Anti-cancer chemotherapy or biologic therapy if administered prior to the first planned dose of study medication (napabucasin or FOLFIRI) within period of time equivalent to the usual cycle length of the regimen. An exception is made for oral fluoropyrimidines (e.g. capecitabine, S-1), where a minimum of 10 days since last dose must be observed prior to the first planned dose of study medication. Standard dose of bevacizumab (5 mg/kg) may be administered prior to FOLFIRI infusion, per Investigator decision, for as long as permanent decision to include or exclude bevacizumab is made prior to patient randomization. Radiotherapy, immunotherapy (including immunotherapy administered for non-malignant diseaseneoplastic treatment purposes), or investigational agents within four weeks of first planned dose of study medication, with the exception of a single dose of radiation up to 8 Gy (equal to 800 RAD) with palliative intent for pain control up to 14 days before randomization.
2. More than one prior chemotherapy regimen administered in the metastatic setting.
3. Major surgery within 4 weeks prior to randomization.
4. Patients with any known brain or leptomeningeal metastases are excluded, even if treated.
5. Women who are pregnant or breastfeeding. Women should not breastfeed while taking study treatment and for 4 weeks after the last dose of napabucasin or while undergoing treatment with FOLFIRI and for 180 days after the last dose of FOLFIRI.
6. Gastrointestinal disorder(s) which, in the opinion of the Qualified/Principal Investigator, would significantly impede the absorption of an oral agent (e.g. intestinal occlusion, active Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection).
7. Unable or unwilling to swallow napabucasin capsules daily.
8. Prior treatment with napabucasin.
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.
10. Known hypersensitivity to 5-fluorouracil/leucovorin
11. Known dihydropyrimidine dehydrogenase (DPD) deficiency
12. Known hypersensitivity to irinotecan
13. Chronic inflammatory bowel disease (Crohn's disease or ulcerative colitis)
14. Patients receiving treatment with St. John's wort or Phenytoin.
15. Patients who plan to receive yellow fever vaccine during the course of the study treatment.
16. Abnormal glucuronidation of bilirubin, known Gilbert's syndrome
17. Patients with QTc interval > 470 milliseconds
18. For patients to be treated with a regimen containing bevacizumab:

    * History of cardiac disease: congestive heart failure (CHF) > New York Heart Association (NYHA) Class II; active coronary artery disease, myocardial infarction within 6 months prior to study entry; unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest) or cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
    * Current uncontrolled hypertension (systolic blood pressure [BP] > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management) as well as prior history of hypertensive crisis or hypertensive encephalopathy.
    * History of arterial thrombotic or embolic events (within 6 months prior to study entry)
    * Significant vascular disease (e.g., aortic aneurysm, aortic dissection, symptomatic peripheral vascular disease)
    * Evidence of bleeding diathesis or clinically significant coagulopathy
    * Major surgical procedure (including open biopsy, significant traumatic injury, etc.) within 28 days, or anticipation of the need for major surgical procedure during the course of the study as well as minor surgical procedure (excluding placement of a vascular access device or bone marrow biopsy) within 7 days prior to study enrollment
    * Proteinuria at screening as demonstrated by urinalysis with proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
    * History of abdominal fistula, gastrointestinal perforation, peptic ulcer, or intra-abdominal abscess within 6 months
    * Ongoing serious, non-healing wound, ulcer, or bone fracture
    * Known hypersensitivity to any component of bevacizumab
    * History of reversible posterior leukoencephalopathy syndrome (RPLS)
    * History of hypersensitivity to Chinese hamster ovary (CHO) cells or other human or humanized recombinant antibodies.
19. Patients with a history of other malignancies except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for > 3 years.
20. Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
21. Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1253 (Actual)
Dates: Start 2016-06; Primary Completion 2020-04-28 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (209):
- United States (74):
  - Alabama Oncology, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - City of Hope- Comprehensive Care Center, Duarte, California
  - University of California-San Diego/Moores UCSD Cancer Center, La Jolla, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Hematology Oncology Santa Monica, Santa Monica, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - St Mary's Hospital & Regional Med Center, Grand Junction, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Florida Cancer Specialists & Research Institute Fort Myers, Fort Myers, Florida
  - Memorial Cancer Institute at Memorial Hospital, Hollywood, Florida
  - Baptist Health Medical Group Oncology, LLC, Miami, Florida
  - Sarah Cannon Research Institution, St. Petersburg, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Suburban Hematology-Oncology Associates, PC - Lawrenceville, Lawrenceville, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Northshore University Healthsystem, Evanston, Illinois
  - Healthcare Research Network III, LLC, Tinley Park, Illinois
  - Northwestern Medicine Cancer Center, Warrenville, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University Health Goshen Center for Cancer Care, Goshen, Indiana
  - Michiana Hematology Oncology, PC, Mishawaka, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Dana Farber, Boston, Massachusetts
  - Umass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Mayo Clinic Arizona, Rochester, Minnesota
  - Research Medical Center, Kansas City, Missouri
  - Missouri Baptist Medical Center ACCRU Network Site, St Louis, Missouri
  - Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Cancer Research Network of Nebraska / Oncology Associates PC, Omaha, Nebraska
  - Tennessee Oncology PLLC, Omaha, Nebraska
  - Darthmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Carol G. Simon Cancer Center, Morristown, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Roswell Park Cancer Center, Buffalo, New York
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Toledo Clinic Cancer Centers, Toledo, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - West Cancer Center, Memphis, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Dallas Center, Dallas, Texas
  - Texas Oncology - Denton South, Denton, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Millenium Oncology, Houston, Texas
  - Texas Health Physicians Group, Plano, Texas
  - Texas Oncology-San Antonio, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology - Wichita Falls Texoma Cancer Center, Wichita Falls, Texas
  - Northern Utah Associates, Ogden, Utah
  - US Oncology - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Virginia Mason, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- Australia (15):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - St Vincent's hospital Melbourne, Fitzroy, New South Wales
  - Port Macquaries Base Hospital, Port Macquarie, New South Wales
  - Northern Cancer Institute, St Leonards, New South Wales
  - Sunshine Coast Hospital and Health Service, Nambour, Queensland
  - Gold Coast University Hosptial, Southport, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Bendigo Hospital, Bendigo, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Western Health, Melbourne, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Prince of Wales Hospital, Randwick
- Belgium (8):
  - Imelda Ziekenhuis, Bonheiden, Antwerpen
  - AZ Turnhout - Campus Sint-Elisabeth, Turnhout, Antwerpen
  - Hôpital Erasme, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi - Site Notre-Dame, Charleroi, Hainaut
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Brussels, Liège
  - UZ Leuven - Campus Gasthuisberg, Leuven, Vlaams Brabant
  - AZ Sint-Jan Brugge - Oostende - Campus Sint-Jan, Bruges, West-Vlaanderen
  - AZ Sint-Lucas - Campus Sint-Lucas, Bruges, West-Vlaanderen
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - University of Toronto - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Saint Michael's Hospital Li Ka Shing Knowledge Institute, Toronto, Ontario
  - St. Mary's Hospital Center, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
- China (3):
  - Beijing Cancer Hospital, Beijing
  - Henan Cancer Hospital, Henan
  - Jiangsu Province Hospital, Jiangsu
- Czechia (4):
  - FN Hradec Kralove, Hradec Králové, Královéhradecký kraj
  - Fakultni nemocnice Brno, Brno
  - Masarykuv onkologicky ustav, Brno
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (11):
  - Centre Paul Papin, Angers
  - Hospitalier Jean Minjoz, Besançon
  - Hôpital Morvan - CHRU de Brest - cancérologie et d'hématolog, Brest
  - CHU Estaing, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer (CLCC), Dijon
  - CHU de Nantes - Hopital Hotel Dieu, Nantes
  - Hôpital Européen Georges Pompidou - Digestive Oncology, Paris
  - Hôpital Privé des Côtes d'Armor - Service oncologie, Plérin
  - Hospital of Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes
  - Centre Rene Gauducheau, Saint-Herblain
- Germany (13):
  - Leopoldina Krankenhaus Med. Klinik 2, Schweinfurt, Bavaria
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Schwerpunkpraxis für Hämatologie und Onkologie, Magdeburg, Saxony-Anhalt
  - Gesundheitszentrum Wetterau, Bad Nauheim
  - Vivantes Klinikum Am Urban, Berlin
  - Charite - Campus Benjamin Franklin (Cbf), Berlin
  - DRK Kliniken Berlin Koepenick, Berlin
  - Charité Universitätsmedizin, Berlin
  - MVZ Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin
  - Facharztzentrum Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Universitätsklinikum Marburg, Marburg
  - Medizinische Universitaetsklin, Ulm
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Israel (9):
  - Ha'Emek Medical Center, Afula
  - The Barzilai Medical Center - Oncology Institute, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Shaare Zedek Medical center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin MC - Oncology, Davidoff Center, Petah Tikva
  - Ziv Medical Center (The Rebecca Sieff Hospital), Safed
  - Tel Aviv Sourasky Medical Center - Oncology, Tel Aviv
  - The Chaim Sheba Medical Centre - Division of Oncology, Tel Litwinsky
- Italy (12):
  - AOU Ospedali Riuniti Umberto I - GM.Lanc, Torrette Di Ancona, Ancona
  - Ospedale Santa Maria del Prato, Feltre, Belluno
  - Irccs Irst, Meldola, Forli
  - AUSL della Romagna, Osp. degli Infermi, Faenza, Ravenna
  - Policlinico S.Orsola Malpighi, AOU di Bologna, Bologna
  - PO di Cremona, ASST di Cremona, Cremona
  - AO S. Martino, IRCCS, IST, Genova
  - Ieo, Irccs, Milan
  - AOU Policlinico di Modena, Modena
  - Università degli studi della Campania "L.Vanvitelli", Napoli
  - Ospedale Guglielmo da Saliceto, AUSL Piacenza, Piacenza
  - AOU Città della Salute e della Scienza di Torino - Molinette, Torino
- Japan (16):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsunami, Ehime
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - ST. Marianna University School of Medicine, Kawasaki, Kanagawa
  - Osaka University Hospital, Suita, Osaka
  - Osaka Medical College Hospital, Takatsuki, Osaka
  - Saitama Cancer Center, Kita-Adachi, Saitama
  - Shizuoka Cancer Center, Sunto, Shizuoka
  - Medical Hospital, Tokyo Medical and Dental University, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The cancer insitute hospital of JFCR (Japanese Foundation For Cancer Research), Koto-ku, Tokyo
  - National Kyushu Cancer Center, Fukuoka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
- Netherlands (5):
  - Medisch Centrum Leeuwarden, Leeuwarden, Provincie Friesland
  - Academisch Medisch Centrum, Amsterdam
  - Spaarne Gasthuis, Hoofddorp
  - Maastricht UMC, Maastricht
  - Elizabeth Tweesteden Ziekenhuis locatie Tilburg, Tilburg
- Singapore (3):
  - National University Cancer Institute, Singapore, Central Singapore
  - National Cancer Centre, Singapore, Central Singapore
  - Raffles Hospital, Singapore, Central Singapore
- South Korea (8):
  - Yeungnam University Medical Center, Daegu, Daegu Gwang'yeogsi
  - National Cancer Centre, Goyang, Gyeonggido
  - Ajou University Hospital, Suwon, Gyeonggido
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'yeogsi
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
- Spain (20):
  - Hospital General Universitario de Elche, Elche, Alicante
  - H.U.V. del Rocío, Seville, Andalusia
  - Hospital Son Llatzer, Baleares, Balearic Islands
  - Institut Català d'Oncologia-Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Complexo Hospital Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario Fundacion Alcorcon (HUFA), Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Consorci Hospital General Universitari Valencia (CHGUV), Comunidad Valenciana, Valencia
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen de la Macarena, Seville
  - H.C.U.Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1253 participants were randomized between October 2016 and March 2019.
Pre-assignment Details: Completers included patients who died, withdrew consent to survival follow up or were lost to follow up.
Groups:
- Napabucasin + FOLFIRI ± Bevacizumab: Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 12 hours (480 mg total daily dose).
  Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will start at least 2 hours following the first daily dose of napabucasin and will be administered every 2 weeks. Irinotecan/leucovorin infusion will follow bevacizumab infusion in selected patients to receive standard dose of bevacizumab (5 mg/kg). Irinotecan 180 mg/m^2 together with leucovorin 400 mg/m^2 will be administered intravenously, over approximately 90 minutes and 2 hours, respectively, starting on Day 1 of Cycle 1, following bevacizumab infusion or at least 2 hours following the first daily dose of napabucasin if bevacizumab is not administered. 5-FU 400 mg/m^2 bolus will be administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m^2/day (total 2400 mg/m^2) continuous infusion. This regimen will be repeated on Day 1 of every 14 day cycle
- FOLFIRI ± Bevacizumab: Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will be administered every 2 weeks. Irinotecan/leucovorin infusion will follow bevacizumab infusion in selected patients to receive standard dose of bevacizumab (5 mg/kg). Irinotecan 180 mg/m^2 together with leucovorin 400 mg/m^2 will be administered intravenously, over approximately 90 minutes and 2 hours, respectively, starting on Day 1 of Cycle 1, following bevacizumab infusion. 5-FU 400 mg/m^2 bolus will be administered intravenously immediately following irinotecan/leucovorin infusion, followed by 5-FU 1200 mg/m^2/day (total 2400 mg/m^2) continuous infusion. This regimen will be repeated on Day 1 of every 14 day cycle.
Period: Overall Study
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
Started | 624 | 629
Discontinued Due to Death | 507 | 499
Completion of Survival Follow-Up Due to Study Completion | 64 | 62
Completed | 571 | 561
Not Completed | 53 | 68
Not completed — Lost to Follow-up | 13 | 11
Not completed — Withdrawal by Subject | 37 | 47
Not completed — Other | 3 | 8
Not completed — Hospice | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab | Total
Number analyzed (Participants) | 624 | 629 | 1253
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (11.17) | 59.6 (11.14) | 59.8 (11.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 254 | 494
  Male | 384 | 375 | 759
Race/Ethnicity, Customized [Number; unit: participants] — Race (White, Black, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Other)
  participants
    White | 375 | 370 | 745
    Black or African American | 29 | 38 | 67
    Asian | 197 | 194 | 391
    American Indian or Alaska Native | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Other | 9 | 12 | 21
    Missing | 13 | 14 | 27
Region of Enrollment [Number; unit: participants] — Region/Country(Australia, Balgium, Canada, China, Czech Republic, France, Germany, Hong Kong, Israel, Italy, Japan, Korea Republic of, Netherlands, Singapore, Spain, United States)
  participants
    Singapore | 8 | 9 | 17
    Hong Kong | 1 | 11 | 12
    United States | 203 | 209 | 412
    Czechia | 18 | 19 | 37
    Japan | 63 | 63 | 126
    Spain | 74 | 62 | 136
    Canada | 21 | 15 | 36
    Netherlands | 16 | 21 | 37
    South Korea | 44 | 39 | 83
    Belgium | 16 | 24 | 40
    China | 62 | 59 | 121
    Italy | 22 | 29 | 51
    Israel | 8 | 10 | 18
    Australia | 36 | 24 | 60
    France | 20 | 21 | 41
    Germany | 12 | 14 | 26
ECOG Performance Status [Count of Participants; unit: Participants] — The ECOG(Eastern Cooperative Oncology Group) Performance Status describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). The higher the score, the more restricted the patient is clinically determined to be.
  Participants
    ECOG: 0 | 333 | 332 | 665
    ECOG: 1 | 291 | 297 | 588

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization until death from any cause.
  Patients who are alive at the time of the interim or the final analyses or who have become lost to follow-up will be censored on the date the patient was last known to be alive.
Time Frame: Randomization to Date of Death from any cause or database cutoff date (28 Apr 2020) (Approximately 43 months)
Population: The pSTAT3 subpopulations will be defined by the results of a Clinical Trial Assay (CTA) for a specimen with an age within a defined cut-section stability (CSS) window.
  A patient with positive pSTAT3 status within a defined CSS window is the one with pSTAT3 positive designated by CTA with specimen age up to 6 months at interim analysis or up to the final CSS window at final analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 624 | 629
months
  Overall Survival (OS), General Population(GP) | 14.29 [13.34 to 15.7] | 13.83 [12.42 to 15.28]
  Overall Survival (OS), ITT-pSTAT3(+): number analyzed (Participants) | 275 | 272
  Overall Survival (OS), ITT-pSTAT3(+) | 13.17 [11.30 to 15.31] | 12.12 [11.24 to 14.06]
Statistical Analysis 1: Comparison: Napabucasin + FOLFIRI ± Bevacizumab vs FOLFIRI ± Bevacizumab; General population; Test type: Superiority; p = 0.3629, Log Rank — 1-sided; Based on stratified log-rank test stratified by actual stratification factors. P-value is nominal p-value without multiplicity adjustment; Hazard Ratio (HR) = 0.976, 95% CI 2-sided [0.854 to 1.117] — Based on Cox Proportional hazards model stratified by actual stratification factors including Time to progression on 1st line therapy, RAS mutation, and Bev as part of study treatment. A HR <1 indicates a lower risk with Arm 1 compared with Arm 2
Statistical Analysis 2: Comparison: Napabucasin + FOLFIRI ± Bevacizumab vs FOLFIRI ± Bevacizumab; activated signal transducers and activators of transcription 3 (pSTAT3)-positive (pSTAT3(+)) Subpopulation patients; Test type: Superiority; p = 0.3782, Log Rank — 1-sided; Based on unstratified log-rank test. P-value is nominal p value without multiplicity adjustment; Hazard Ratio (HR) = 0.969, 95% CI 2-sided [0.797 to 1.179] — Hazard Ratio is for Napabucasin + FOLFIRI ± bev vs FOLFIRI ± bev. Based on unstratified Cox proportional hazards model. A hazard ratio <1 indicates a lower risk with Napabucasin+ FOLFIRI ± bev compared with FOLFIRI ± bev

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first objective documentation of disease progression per RECIST 1.1 (PD) or death, whichever comes first.
Time Frame: Randomization to Date of Death or until the date of first documented objective disease progression or database cutoff date (28 Apr 2020) (Approximately 43 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 624 | 629
months
  Progression-Free Survival (PFS), General Population(GP) | 5.55 [5.39 to 5.78] | 5.62 [5.45 to 6.34]
  Progression-Free Survival (PFS) , ITT-pSTAT3(+): number analyzed (Participants) | 275 | 272
  Progression-Free Survival (PFS) , ITT-pSTAT3(+) | 5.39 [4.14 to 5.62] | 5.55 [4.44 to 5.91]
Statistical Analysis 1: Comparison: Napabucasin + FOLFIRI ± Bevacizumab vs FOLFIRI ± Bevacizumab; General population; Test type: Superiority; p = 0.7307, Log Rank — 1-sided; Based on stratified log rank test stratified by actual stratification factors . P-value is nominal p-value without multiplicity adjustment; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.917 to 1.180] — Based on Cox Proportional hazards model stratified by actual stratification . A HR <1 indicates a lower risk with Arm 1 compared with Arm 2
Statistical Analysis 2: Comparison: Napabucasin + FOLFIRI ± Bevacizumab vs FOLFIRI ± Bevacizumab; activated signal transducers and activators of transcription 3 (pSTAT3)-positive (pSTAT3(+)) Subpopulation patients; Test type: Superiority; p = 0.7434, Log Rank — 1-sided; Based on unstratified log-rank test. P-value is nominal p-value without multiplicity adjustment; Hazard Ratio (HR) = 1.064, 95% CI 2-sided [0.883 to 1.283] — Hazard ratio is for Napabucasin + FOLFIRI ± bev vs FOLFIRI ± bev. Based on unstratified Cox Proportional hazards model. A hazard ratio <1 indicates a lower risk with Napabucasin + FOLFIRI ± bev compared with FOLFIRI ± bev

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1. The primary estimate of DCR will be based on patients with measurable disease by RECIST 1.1 at randomization
Time Frame: as for outcome 2
Population: Analysis population of DCR will be based on patients with measurable disease by RECIST 1.1 at randomization. A patient with positive pSTAT3 status within a defined CSS window is the one with pSTAT3 positive designated by CTA with specimen age up to 6 months at interim analysis or up to the final CSS window at final analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Napabucasin + FOLFIRI ± Bevacizumab: Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 12 hours (480 mg total daily dose).
  Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will start at least 2 hours following the first daily dose of napabucasin and will be administered every 2 weeks. This regimen will be repeated on Day 1 of every 14 day cycle. Analysis population of DCR will be based on patients with measurable disease by RECIST 1.1 at randomization.
- FOLFIRI ± Bevacizumab: Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will be administered every 2 weeks. This regimen will be repeated on Day 1 of every 14 day cycle. Analysis population of DCR will be based on patients with measurable disease by RECIST 1.1 at randomization.
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 593 | 609
percentage of participants
  Disease Control Rate (DCR), General Population(GP) | 69.6 [65.8 to 73.3] | 69.1 [65.3 to 72.8]
  Disease Control Rate (DCR), ITT-pSTAT3(+): number analyzed (Participants) | 268 | 266
  Disease Control Rate (DCR), ITT-pSTAT3(+) | 67.2 [61.2 to 72.8] | 70.3 [64.4 to 75.7]
Statistical Analysis 1: Comparison: Napabucasin + FOLFIRI ± Bevacizumab vs FOLFIRI ± Bevacizumab; General population; Test type: Superiority; p = 0.4797, Cochran-Mantel-Haenszel — 1-sided; Based on Cochran-Mantel-Haenszel test stratified by actual stratification factors. P-value is nominal p-value without multiplicity adjustment; rate difference = 0.1, 95% CI 2-sided [-4.9 to 5.2] — Treatment difference and 95% CI is based on Harmonic Means method adjusting stratification factor
Statistical Analysis 2: Comparison: Napabucasin + FOLFIRI ± Bevacizumab vs FOLFIRI ± Bevacizumab; activated signal transducers and activators of transcription 3 (pSTAT3)-positive (pSTAT3(+)) Subpopulation patients; Test type: Superiority; p = 0.783, Z test — 1-sided; Based on one-sided Z test. P-value is nominal p-value without multiplicity adjustment; rate difference = -3.1, 95% CI 2-sided [-11.0 to 4.7] — Treatment difference and 95% CI is based on normal approximation method

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the proportion of patients with a documented complete response and partial response (CR + PR) based on RECIST 1.1. The primary estimate for ORR will be based on patients with measurable disease by RECIST 1.1 at randomization.
Time Frame: as for outcome 2
Population: Analysis set for ORR will be based on patients with measurable disease by RECIST 1.1 at randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Napabucasin + FOLFIRI ± Bevacizumab: Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 12 hours (480 mg total daily dose).
  Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will start at least 2 hours following the first daily dose of napabucasin and will be administered every 2 weeks. This regimen will be repeated on Day 1 of every 14 day cycle. Analysis set for ORR will be based on patients with measurable disease by RECIST 1.1 at randomization.
- FOLFIRI ± Bevacizumab: Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will be administered every 2 weeks. This regimen will be repeated on Day 1 of every 14 day cycle. Analysis set for ORR will be based on patients with measurable disease by RECIST 1.1 at randomization.
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 593 | 609
percentage of participants
  Objective Response Rate (ORR), General Population(GP) | 13.8 [11.2 to 16.9] | 14.6 [11.9 to 17.7]
  Objective Response Rate (ORR), ITT-pSTAT3(+): number analyzed (Participants) | 268 | 266
  Objective Response Rate (ORR), ITT-pSTAT3(+) | 11.9 [8.3 to 16.4] | 13.9 [10.0 to 18.7]
Statistical Analysis 1: Comparison: Napabucasin + FOLFIRI ± Bevacizumab vs FOLFIRI ± Bevacizumab; General population; Test type: Superiority; p = 0.6776, Cochran-Mantel-Haenszel — 1-sided; Based on Cochran-Mantel-Haenszel test stratified by actual stratification factors. P-value is nominal p-value without multiplicity adjustment; rate difference = -0.9, 95% CI 2-sided [-4.8 to 3.0] — Treatment difference and 95% CI is based on Harmonic Means method adjusting stratification factor
Statistical Analysis 2: Comparison: Napabucasin + FOLFIRI ± Bevacizumab vs FOLFIRI ± Bevacizumab; activated signal transducers and activators of transcription 3 (pSTAT3)-positive (pSTAT3(+)) Subpopulation patients; Test type: Superiority; p = 0.7513, Z test — 1-sided; Based on one-sided Z test. P-value is nominal p-value without multiplicity adjustment; rate difference = -2.0, 95% CI 2-sided [-7.7 to 3.7] — Treatment difference and 95% CI is based on normal approximation method

5. Secondary Outcome: Mean Change From Baseline for Global Health Status at Time 2 (Cycle 5 Day 1) and Time 4 (Cycle 9 Day 1).
Description: The Quality of Life (QoL) of patients will be assessed using European Organization for Research and Treatment of Cancer Quality of Life questionnaire (EORTC-QLQ-C30) (EORTC QLQ-30) while the patient remains on study treatment (FOLFIRI with or without BBI-608). EORTC QLQ-30 is used to assess the overall quality of life in cancer patients using 28 questions with a 4 point scale. (1 'Not at all' to 4'Very Much'); 2 questions use a 7-point sale (1 'Very Poor' to 7 'Excellent'). Scores are averaged and transformed to 0-100 scale; higher overall score = better quality of life.
Time Frame: From baseline at Time 2 (Cycle 5 Day 1), approximately 57 days and Time 4 (Cycle 9 Day 1), approximately 113 days
Population: The number of patients is with at least one valid assessment at each analysis window
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Napabucasin + FOLFIRI ± Bevacizumab: Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 12 hours (480 mg total daily dose).
  Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will start at least 2 hours following the first daily dose of napabucasin and will be administered every 2 weeks. This regimen will be repeated on Day 1 of every 14 day cycle. Number of patients is with at least one valid assessment at each analysis window.
- FOLFIRI ± Bevacizumab: Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will be administered every 2 weeks. This regimen will be repeated on Day 1 of every 14 day cycle. Number of patients is with at least one valid assessment at each analysis window.
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 622 | 626
score on a scale
  Mean Change From Baseline for Global Health status at Time 2 (Cycle 5 Day 1). General Population: number analyzed (Participants) | 376 | 341
  Mean Change From Baseline for Global Health status at Time 2 (Cycle 5 Day 1). General Population | -7.07 (21.936) | -5.45 (20.607)
  Mean Change From Baseline for Global Health status at Time 4 (Cycle 9 Day 1). General Population: number analyzed (Participants) | 370 | 360
  Mean Change From Baseline for Global Health status at Time 4 (Cycle 9 Day 1). General Population | -7.70 (21.932) | -5.58 (21.590)

6. Secondary Outcome: Mean Change From Baseline for Physical Functioning Status at Time 2 (Cycle 5 Day 1) and Time 4 (Cycle 9 Day 1).
Description: as for outcome 5
Time Frame: From baseline at Time 2 (Cycle 5 Day 1) and Time 4 (Cycle 9 Day 1)
Population: The number of patients is with at least one valid assessment at each analysis window.
Measure: Mean (Standard Deviation); unit: QOL score on a scale
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 622 | 626
QOL score on a scale
  Mean Change From Baseline for Physical Functioning at Time 2 (Cycle 5 Day 1). General Population: number analyzed (Participants) | 375 | 343
  Mean Change From Baseline for Physical Functioning at Time 2 (Cycle 5 Day 1). General Population | -5.86 (17.204) | -3.94 (14.472)
  Mean Change From Baseline for Physical Functioning at Time 4 (Cycle 9 Day 1). General Population: number analyzed (Participants) | 369 | 363
  Mean Change From Baseline for Physical Functioning at Time 4 (Cycle 9 Day 1). General Population | -6.37 (15.095) | -4.22 (15.023)

7. Secondary Outcome: Number of Patients With Adverse Events in the General Population
Description: All patients who have received at least one dose of either BBI-608 or FOLFIRI will be included in the safety analysis according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE) version 4.0. The incidence of adverse events will be summarized by type of adverse event and severity.
Time Frame: All adverse event are collected from date of signed informed consent until 30 days after protocol treatment discontinuation. Outcome followed until study discontinuation up to 4 years
Population: All patients who received at least 1 dose of study drug (BBI-608 and/or FOLFIRI) with treatment assignment designated according to the actual study treatment received. Adverse event is analyzed in the SAS population.
Measure: Count of Participants; unit: Participants
Groups:
- Napabucasin + FOLFIRI ± Bevacizumab: All patients who received at least 1 dose of study drug (BBI-608 and/or FOLFIRI) with treatment assignment designated according to the actual study treatment received. Napabucasin 240 mg will be administered orally, twice daily, with doses separated by approximately 12 hours (480 mg total daily dose).
  Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will start at least 2 hours following the first daily dose of napabucasin and will be administered every 2 weeks. Irinotecan/leucovorin infusion will follow bevacizumab infusion in selected patients to receive standard dose of bevacizumab (5 mg/kg). This regimen will be repeated on Day 1 of every 14 day cycle.
- FOLFIRI ± Bevacizumab: All patients who received at least 1 dose of study drug (FOLFIRI) with treatment assignment designated according to the actual study treatment received. Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will be administered every 2 weeks. Irinotecan/leucovorin infusion will follow bevacizumab infusion in selected patients to receive standard dose of bevacizumab (5 mg/kg). This regimen will be repeated on Day 1 of every 14 day cycle.
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
Number analyzed (Participants) | 622 | 610
Participants
  Number of Patients with Adverse Events in the General Population | 619 | 602
  Number of Patients with Adverse Events in the pSTAT3(+) Subpopulation: number analyzed (Participants) | 275 | 269
  Number of Patients with Adverse Events in the pSTAT3(+) Subpopulation | 275 | 266

ADVERSE EVENTS:
Time Frame: All adverse event are collected from date of signed informed consent until 30 days after protocol treatment discontinuation. Outcome followed until study discontinuation.
Description: All adverse event are collected from date of signed informed consent until 30 days after protocol treatment discontinuation. Outcome followed until study discontinuation up to 4 years.
  All cause mortality is analyzed in the ITT population. That's why total number of participants at risk in the ITT population (624 Arm A, 629 Arm B) appears inconsistent with total number of participants at risk in the adverse event analysis in the SAS population (622 Arm A, 610 Arm B)
Groups:
- FOLFIRI ± Bevacizumab: All patients who received at least 1 dose of study drug (BBI-608 and/or FOLFIRI) with treatment assignment designated according to the actual study treatment received. Addition of bevacizumab to the FOLFIRI regimen will be permissible. FOLFIRI chemotherapy infusion will be administered every 2 weeks. Irinotecan/leucovorin infusion will follow bevacizumab infusion in selected patients to receive standard dose of bevacizumab (5 mg/kg). This regimen will be repeated on Day 1 of every 14 day cycle.
Arm/Group | Napabucasin + FOLFIRI ± Bevacizumab | FOLFIRI ± Bevacizumab
All-Cause Mortality (participants affected / at risk) | 507/624 | 499/629
Serious Adverse Events (participants affected / at risk) | 234/622 | 201/610
Other Adverse Events (participants affected / at risk) | 619/622 | 602/610
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin + FOLFIRI ± Bevacizumab (N=622) | FOLFIRI ± Bevacizumab (N=610)
Diarrhoea (Gastrointestinal disorders) | 39 | 19
Abdominal Pain (Gastrointestinal disorders) | 17 | 16
Intestinal Obstruction (Gastrointestinal disorders) | 10 | 15
Small Intestinal Obstruction (Gastrointestinal disorders) | 10 | 12
Vomiting (Gastrointestinal disorders) | 10 | 8
Nausea (Gastrointestinal disorders) | 9 | 4
Ileus (Gastrointestinal disorders) | 4 | 8
Ascites (Gastrointestinal disorders) | 3 | 3
Intestinal Perforation (Gastrointestinal disorders) | 3 | 2
Large Intestinal Obstruction (Gastrointestinal disorders) | 3 | 4
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 2 | 3
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 1
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 2 | 1
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 1 | 0
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Toxicity (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 1 | 0
Large Intestinal Stenosis (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Obstruction Gastric (Gastrointestinal disorders) | 1 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenal Perforation (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1
Pneumatosis Intestinalis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 18 | 16
Disease Progression (General disorders) | 17 | 15
General Physical Health Deterioration (General disorders) | 5 | 5
Asthenia (General disorders) | 4 | 4
Fatigue (General disorders) | 4 | 2
Death (General disorders) | 2 | 1
Mucosal Inflammation (General disorders) | 2 | 1
Non-Cardiac Chest Pain (General disorders) | 2 | 1
Chills (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Mucosal Toxicity (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 2
Pain (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 7 | 10
Urinary Tract Infection (Infections and infestations) | 6 | 0
Pneumonia (Infections and infestations) | 4 | 8
Anal Abscess (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 2 | 2
Clostridium Difficile Colitis (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 2 | 1
Abdominal Infection (Infections and infestations) | 1 | 0
Abdominal Sepsis (Infections and infestations) | 1 | 0
Appendicitis Perforated (Infections and infestations) | 1 | 0
Bacterial Sepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Colonic Abscess (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Enterocolitis Infectious (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Infected Dermal Cyst (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Nosocomial Infection (Infections and infestations) | 1 | 0
Perirectal Abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 1
Peritonsillar Abscess (Infections and infestations) | 1 | 0
Pneumonia Influenzal (Infections and infestations) | 1 | 0
Pseudomonas Bronchitis (Infections and infestations) | 1 | 0
Rectal Abscess (Infections and infestations) | 1 | 0
Retroperitoneal Abscess (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 4
Urinary Tract Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 1
Viral Infection (Infections and infestations) | 1 | 0
Abdominal Abscess (Infections and infestations) | 0 | 1
Abdominal Wall Abscess (Infections and infestations) | 0 | 1
Abscess Jaw (Infections and infestations) | 0 | 1
Abscess Rupture (Infections and infestations) | 0 | 1
Anorectal Infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Coccidioidomycosis (Infections and infestations) | 0 | 1
Community Acquired (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Fungal Sepsis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 0 | 1
Ophthalmic Herpes Zoster (Infections and infestations) | 0 | 1
Pelvic Abscess (Infections and infestations) | 0 | 1
Pelvic Infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1
Psoas Abscess (Infections and infestations) | 0 | 1
Pulmonary Sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 4
Pyonephrosis (Infections and infestations) | 0 | 1
Respiratory Tract (Infections and infestations) | 0 | 1
Streptococcal Bacteraemia (Infections and infestations) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 15 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 4 | 3
Failure To Thrive (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 9 | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 8 | 12
Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 1
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 2 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 2 | 0
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 2 | 3
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 | 1
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Stoma Complication (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hypotension (Vascular disorders) | 6 | 3
Deep Vein Thrombosis (Vascular disorders) | 2 | 2
Embolism (Vascular disorders) | 2 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypovolaemic Shock (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 1
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 2 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Gallbladder Necrosis (Hepatobiliary disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Jaundice Cholestatic (Hepatobiliary disorders) | 1 | 1
Bile Duct Stenosis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Liver Injury (Hepatobiliary disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 7 | 3
Acute Prerenal Failure (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Prerenal Failure (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Hydroureter (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 2
Urinary Tract Obstruction (Renal and urinary disorders) | 0 | 2
Atrial Fibrillation (Cardiac disorders) | 3 | 4
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 1 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Blood Bilirubin Increased (Investigations) | 2 | 1
Neutrophil Count Decreased (Investigations) | 2 | 8
Platelet Count Decreased (Investigations) | 2 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Myocardial Necrosis Marker Increased (Investigations) | 1 | 0
Red Blood Cell Count Decreased (Investigations) | 1 | 0
Blood Uric Acid Increased (Investigations) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 2
Syncope (Nervous system disorders) | 2 | 3
Altered State Of Consciousness (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0
Superior Sagittal Sinus Thrombosis (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Spinal Cord Disorder (Nervous system disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Fracture Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases To Kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional State (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Device Dislocation (Product Issues) | 1 | 0
Thrombosis In Device (Product Issues) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 2
Tumour Excision (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin + FOLFIRI ± Bevacizumab (N=622) | FOLFIRI ± Bevacizumab (N=610)
Anaemia (Blood and lymphatic system disorders) | 154 | 148
Neutropenia (Blood and lymphatic system disorders) | 154 | 165
Thrombocytopenia (Blood and lymphatic system disorders) | 36 | 24
Leukopenia (Blood and lymphatic system disorders) | 32 | 43
Diarrhoea (Gastrointestinal disorders) | 526 | 329
Nausea (Gastrointestinal disorders) | 376 | 308
Vomiting (Gastrointestinal disorders) | 256 | 180
Abdominal Pain (Gastrointestinal disorders) | 255 | 154
Constipation (Gastrointestinal disorders) | 126 | 173
Stomatitis (Gastrointestinal disorders) | 92 | 118
Abdominal Pain Upper (Gastrointestinal disorders) | 63 | 46
Dyspepsia (Gastrointestinal disorders) | 56 | 39
Proctalgia (Gastrointestinal disorders) | 35 | 20
Abdominal Distension (Gastrointestinal disorders) | 34 | 31
Fatigue (General disorders) | 235 | 219
Asthenia (General disorders) | 135 | 119
Pyrexia (General disorders) | 117 | 100
Mucosal Inflammation (General disorders) | 60 | 90
Oedema Peripheral (General disorders) | 45 | 48
Malaise (General disorders) | 43 | 34
Urinary Tract Infection (Infections and infestations) | 71 | 40
Upper Respiratory Tract Infection (Infections and infestations) | 44 | 43
Neutrophil Count Decreased (Investigations) | 149 | 179
Weight Decreased (Investigations) | 106 | 54
White Blood Cell Count Decreased (Investigations) | 87 | 109
Aspartate Aminotransferase Increased (Investigations) | 75 | 67
Alanine Aminotransferase Increased (Investigations) | 67 | 57
Blood Alkaline Phosphatase Increased (Investigations) | 59 | 35
Platelet Count Decreased (Investigations) | 42 | 47
Blood Bilirubin Increased (Investigations) | 30 | 32
Decreased Appetite (Metabolism and nutrition disorders) | 233 | 189
Hypokalaemia (Metabolism and nutrition disorders) | 103 | 57
Dehydration (Metabolism and nutrition disorders) | 57 | 36
Hypoalbuminaemia (Metabolism and nutrition disorders) | 33 | 29
Back Pain (Musculoskeletal and connective tissue disorders) | 75 | 84
Headache (Nervous system disorders) | 85 | 73
Dizziness (Nervous system disorders) | 59 | 47
Dysgeusia (Nervous system disorders) | 46 | 59
Neuropathy Peripheral (Nervous system disorders) | 32 | 22
Cholinergic Syndrome (Nervous system disorders) | 20 | 33
Insomnia (Psychiatric disorders) | 54 | 84
Chromaturia (Renal and urinary disorders) | 70 | 4
Proteinuria (Renal and urinary disorders) | 54 | 44
Cough (Respiratory, thoracic and mediastinal disorders) | 72 | 75
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 60 | 79
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57 | 46
Hiccups (Respiratory, thoracic and mediastinal disorders) | 41 | 29
Alopecia (Skin and subcutaneous tissue disorders) | 133 | 159
Rash (Skin and subcutaneous tissue disorders) | 31 | 41
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 30 | 33
Hypertension (Vascular disorders) | 58 | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT02753127/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT02753127/SAP_001.pdf